CLINICAL TRIAL: NCT04098055
Title: Effectiveness of Custom-made Foot Orthoses in Patients With Systemic Lupus Erythematous
Brief Title: Effect of Insoles in Patients With Systemic Lupus Erythematosus
Acronym: EISLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Pedro V. Munuera-Martínez, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SLE
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lupus Erythematosus, Systemic; Foot Orthoses; Musculoskeletal Pain
Keywords: Lupus Erythematosus, Systemic; Foot Orthoses; Foot; Pain
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Musculoskeletal Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made foot orthoses (Experimental)
  Interventions: Device: Custom-Made Foot Orthoses
- Control Group (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Custom-Made Foot Orthoses — The foot orthoses were custom made using phenolic foam molds of the feet. They consisted of a polypropylene layer of 2 mm from heel to just proximal to the metatarsal heads, an upper sheet of 30 Shore A polyethylene foam.
  Arms: Custom-made foot orthoses
Device: Placebo — The insole made using phenolic foam molds of the feet. They consisted of an upper sheet of 30 Shore A polyethylene foam.
  Arms: Control Group

SUMMARY:
Demonstrate that custom-made insoles improve painful symptomatology, health and foot function in subjects with SLE and podiatric involvement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more.
* Medical diagnosis of LES.
* Foot involvement.

Exclusion Criteria:

* Treatment with foot orthoses.
* LES with acute symptomatic flare.
* Ulcers.
* Skin involvement.
* Neurological problems.
* Cognitive deterioration.
* Need for walking assistance.
* Refused to change footwear to use the foot orthoses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
11-point Numeric Pain Rating Scale | 1 minute
  With a range of 0 = no pain to 10 = pain as bad as it can be.
SF- 12 Quality of Life | 10 minutes
  To describe the relationships among functional health status measures. This has values between 0 and 100, with higher values corresponding to lower quality of life.
Foot Function | 5 minutes
  Foot Function Index
Foot Disability | 5 minutes
  Manchester Foot Pain and Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Podiatry, Seville, Spain

REFERENCES:
- [Result] Pipili C, Sfritzeri A, Cholongitas E. Deforming arthropathy in systemic lupus erythematosus. Eur J Intern Med. 2008 Nov;19(7):482-7. doi: 10.1016/j.ejim.2008.01.017. Epub 2008 Apr 1. PMID 19013374
- [Result] Otter SJ, Kumar S, Gow P, Dalbeth N, Corkill M, Rohan M, Davies KA, Pankathelam S, Rome K. Patterns of foot complaints in systemic lupus erythematosus: a cross sectional survey. J Foot Ankle Res. 2016 Mar 22;9:10. doi: 10.1186/s13047-016-0143-8. eCollection 2016. PMID 27006702
- [Result] Reina-Bueno M, Vazquez-Bautista MDC, Perez-Garcia S, Rosende-Bautista C, Saez-Diaz A, Munuera-Martinez PV. Effectiveness of custom-made foot orthoses in patients with rheumatoid arthritis: a randomized controlled trial. Clin Rehabil. 2019 Apr;33(4):661-669. doi: 10.1177/0269215518819118. Epub 2018 Dec 17. PMID 30556429
- [Derived] Reina-Bueno M, Vazquez-Bautista MDC, Palomo-Toucedo IC, Dominguez-Maldonado G, Castillo-Lopez JM, Ramos-Ortega J, Munuera-Martinez PV. Effectiveness of custom-made foot orthoses in patients with systemic lupus erythaematosus: protocol for a randomised controlled trial. BMJ Open. 2021 Mar 1;11(3):e042627. doi: 10.1136/bmjopen-2020-042627. PMID 33649056